CLINICAL TRIAL: NCT02689804
Title: Pharmacokinetics of Levonorgestrel and Ulipristal Acetate Emergency Contraception in Women With Normal and Obese Body Mass Index
Brief Title: EC PK in Women With Normal and Obese BMI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Carolyn L. Westhoff, Director, Division of Family Planning and Preventive Services, Columbia University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: AAAP1857
Record Dates: First submitted 2016-02-16; First posted 2016-02-24 (Estimated); Results first posted 2017-07-07 (Actual); Last update posted 2017-07-07 (Actual); Status verified 2017-06

CONDITIONS: Contraception
Keywords: Emergency contraception
MeSH Terms: interventions — Levonorgestrel; Contraceptives, Postcoital; ulipristal acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Normal-BMI (Other): Women with normal BMI will receive the first emergency contraception (EC) dose and complete pharmacokinetics (PK) assessments; then return to the clinic after at least 8 days to receive the second study drug and complete the same assessments. The study drugs Levonorgestrel (LNG-EC) and Ulipristal Acetate (UPA-EC) will be given in random order.
  Interventions: Drug: LNG-EC; Drug: UPA-EC
- Obese-BMI (Other): Women with obese BMI will receive the first emergency contraception (EC) dose and complete pharmacokinetics (PK) assessments; then return to the clinic after at least 8 days to receive the second study drug and complete the same assessments. The study drugs Levonorgestrel (LNG-EC) and Ulipristal Acetate (UPA-EC) will be given in random order.
  Interventions: Drug: LNG-EC; Drug: UPA-EC

INTERVENTIONS:
Drug: LNG-EC — FDA-approved emergency contraceptive pill containing levonorgestrel 1.5mg
  Other Names: Levonorgestrel (LNG) emergency contraceptive (EC); Next Choice One Dose
Drug: UPA-EC — FDA-approved emergency contraceptive pill containing ulipristal acetate 30mg
  Other Names: Ulipristal acetate (UPA) emergency contraceptive (EC); ella

SUMMARY:
A well-designed pharmacokinetics (PK) study may identify the physiologic basis for observed differences in levonorgestrel emergency contraception (LNG-EC) and ulipristal acetate emergency contraception (UPA-EC) failure rates in women with normal and obese BMI. The investigators propose a study to compare serum LNG and UPA levels after administration of a single-dose of LNG-EC or UPA-EC. The investigators hypothesize that there will be no difference in PK parameters between women with normal BMI and obese women.

DETAILED DESCRIPTION:
Eligible women will present to the division research office, at which time a history and physical exam will be completed. Each participant's BMI will be confirmed and she will be assigned to one of two BMI groups (18.5-24.9 versus 30-39.9). At the conclusion of the enrollment visit, the research coordinator will randomize each woman to receive a single-dose pill of either levonorgestrel 1.5mg (like Plan B One-Step® or its generic formulations) or ulipristal acetate 30mg (ellaOne®) on two separate occasions.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-45 years
* English-speaking
* BMI 18.5-24.9 kg/m2 or obese BMI 30.0-39.9 kg/m2
* Regular menstrual cycles
* No use of medroxyprogesterone acetate at least 6 months prior to study enrollment, unless resumption of two menstrual cycles
* No use of levonorgestrel intrauterine system (levonorgestrel-IUS), etonogestrel implant or combined hormonal contraception at least one month prior to the study and resumption of one menstrual cycle
* Women who are postpartum or post-abortion will be included if they have had at least one menstrual cycle since their last pregnancy

Exclusion Criteria:

* Prior allergic reaction to LNG-EC or UPA-EC
* Use of hormonal emergency contraception within the past month
* Women who are currently pregnant or who are currently breastfeeding
* History of cancer other than non-melanoma skin cancer
* Medical or surgical conditions or conditions requiring therapies known to impact sex steroid production or metabolism

  * Use of HAART therapy for management of HIV infection
  * Concomitant use of CYP3A4 inducers like rifampin, barbiturates, carbamazepine, lamotrigine, bosentan, felbamate, griseofulvin, oxcarbazepine, phenytoin, St. John's Wort and topiramate
* Current participation in any other trial of an investigational medicine or device in the three months leading up to this study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2015-07-10 (Actual); Primary Completion 2015-12-29 (Actual); Study Completion 2017-02-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn L Westhoff, MD, Principal Investigator — Director, Division of Family Planning and Preventive Services; Piyapa Praditpan, MD, Study Director — Clinical instructor, Division of Family Planning and Preventive Services
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Glasier A, Cameron ST, Blithe D, Scherrer B, Mathe H, Levy D, Gainer E, Ulmann A. Can we identify women at risk of pregnancy despite using emergency contraception? Data from randomized trials of ulipristal acetate and levonorgestrel. Contraception. 2011 Oct;84(4):363-7. doi: 10.1016/j.contraception.2011.02.009. Epub 2011 Apr 2. PMID 21920190
- [Background] Kapp N, Abitbol JL, Mathe H, Scherrer B, Guillard H, Gainer E, Ulmann A. Effect of body weight and BMI on the efficacy of levonorgestrel emergency contraception. Contraception. 2015 Feb;91(2):97-104. doi: 10.1016/j.contraception.2014.11.001. Epub 2014 Nov 8. PMID 25528415
- [Background] Gemzell-Danielsson K, Kardos L, von Hertzen H. Impact of bodyweight/body mass index on the effectiveness of emergency contraception with levonorgestrel: a pooled-analysis of three randomized controlled trials. Curr Med Res Opin. 2015 Dec;31(12):2241-8. doi: 10.1185/03007995.2015.1094455. Epub 2015 Oct 27. PMID 26368848
- Available data/document: Publication — http://dx.doi.org/10.1016/j.contraception.2017.01.004 — Results Reference: Yes

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No significant events in the study that occur after participant enrollment, but prior to assignment of participants to an arm or group.
Groups:
- Obese-MRI: Women with obese BMI will receive the first emergency contraception (EC) dose and complete pharmacokinetics (PK) assessments; then return to the clinic after at least 8 days to receive the second study drug and complete the same assessments. The study drugs Levonorgestrel (LNG-EC) and Ulipristal Acetate (UPA-EC) will be given in random order.
Period: Overall Study
Arm/Group | Normal-BMI | Obese-MRI
Started | 18 | 16
Completed | 16 | 16
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Population: This is a cross-over study with the same 32 participants receiving each study drug. 34 participants were enrolled into this study but 2 participants discontinued. The final sample includes a total of 16 normal-BMI women and 16 obese-BMI women.
Groups:
- Normal-BMI: Women with normal BMI will receive the first EC dose and complete PK assessments; then return to the clinic after at least 8 days to receive the second study drug and complete the same assessments. The study drugs (LNG-EC and UPA-EC will be given in random order).
- Obese-BMI: Women with obese BMI will receive the first EC dose and complete PK assessments; then return to the clinic after at least 8 days to receive the second study drug and complete the same assessments. The study drugs (LNG-EC and UPA-EC will be given in random order).
- Total: Total of all reporting groups
Arm/Group | Normal-BMI | Obese-BMI | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Continuous [Mean (Full Range); unit: years] | 28.8 [19 to 35] | 32.3 [21 to 45] | 30 [19 to 45]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 16 | 32
  Male | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16 | 16 | 32

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve From Time 0 to 24 Hours of Serum LNG Concentration
Description: LNG-EC PK parameter (AUC 0-24 h) in women with normal and obese BMI women.
Time Frame: Up to 24 hours
Population: Cross-over study: 16 normal-BMI and 16 obese-BMI enrolled and each participant received both drugs in random order.
Measure: Mean (Inter-Quartile Range); unit: ng*h/mL
Groups:
- Normal-BMI: Women with normal BMI will receive the first EC dose and complete PK assessments; then return to the clinic after at least 8 days to receive the second study drug and complete the same assessments. The study drugs LNG-EC and UPA-EC will be given in random order.
- Obese-BMI: Women with obese BMI will receive the first EC dose and complete PK assessments; then return to the clinic after at least 8 days to receive the second study drug and complete the same assessments. The study drugs LNG-EC and UPA-EC will be given in random order.
Arm/Group | Normal-BMI | Obese-BMI
Number analyzed (Participants) | 16 | 16
ng*h/mL | 208.5 [171.4 to 245.6] | 100.8 [82.9 to 118.7]
Statistical Analysis 1: Comparison: Normal-BMI vs Obese-BMI; Test type: Superiority; p < 0.01, t-test, 2 sided

2. Primary Outcome: Area Under the Curve From Time 0 to 24 Hours of Serum UPA Concentration
Description: UPA-EC PK parameter (AUC 0-24 h) in women with normal and obese BMI women.
Time Frame: Up to 24 hours
Population: Cross-over study: 16 normal-BMI and 16 obese-BMI enrolled and each participant received both drugs in random order.
Measure: Mean (Inter-Quartile Range); unit: ng*h/mL
Arm/Group | Normal-BMI | Obese-BMI
Number analyzed (Participants) | 16 | 16
ng*h/mL | 293.5 [237.3 to 349.8] | 362.5 [230.9 to 494.1]
Statistical Analysis 1: Comparison: Normal-BMI vs Obese-BMI; Test type: Superiority; p = 0.15, t-test, 2 sided

3. Secondary Outcome: Elimination Half-life of Serum LNG
Description: (t1/2) calculated in women with normal and obese BMI
Time Frame: Up to 24 hours
Population: Cross-over study: 16 normal-BMI and 16 obese-BMI enrolled and each participant received both drugs in random order.
Measure: Mean (Inter-Quartile Range); unit: h
Arm/Group | Normal-BMI | Obese-BMI
Number analyzed (Participants) | 16 | 16
h | 27.0 [22.2 to 31.8] | 50.4 [44.6 to 56.3]

4. Secondary Outcome: Elimination Half-life of Serum UPA
Description: (t1/2) calculated in women with normal and obese BMI
Time Frame: Up to 24 hours
Population: Cross-over study: 16 normal-BMI and 16 obese-BMI enrolled and each participant received both drugs in random order.
Measure: Mean (Inter-Quartile Range); unit: h
Groups:
- Obese-MRI: Women with obese BMI will receive the first EC dose and complete PK assessments; then return to the clinic after at least 8 days to receive the second study drug and complete the same assessments. The study drugs LNG-EC and UPA-EC will be given in random order.
Arm/Group | Normal-BMI | Obese-MRI
Number analyzed (Participants) | 16 | 16
h | 34.9 [24.0 to 45.8] | 65.9 [50.8 to 81.0]

5. Secondary Outcome: Clearance of Serum LNG
Description: (Cl) calculated in women with normal and obese BMI
Time Frame: Up to 24 hours
Measure: Mean (Inter-Quartile Range); unit: L/h
Arm/Group | Normal-BMI | Obese-MRI
Number analyzed (Participants) | 16 | 16
L/h | 4.8 [3.8 to 5.8] | 9.8 [8.3 to 11.3]

6. Secondary Outcome: Clearance of Serum UPA
Description: (Cl) calculated in women with normal and obese BMI
Time Frame: Up to 24 hours
Measure: Mean (Inter-Quartile Range); unit: L/h
Arm/Group | Normal-BMI | Obese-MRI
Number analyzed (Participants) | 16 | 16
L/h | 4.1 [3.2 to 5.0] | 3.0 [1.8 to 4.2]

7. Secondary Outcome: Maximum Concentration of Serum LNG
Description: (Cmax) calculated in women with normal and obese BMI
Time Frame: Up to 24 hours
Measure: Mean (Inter-Quartile Range); unit: ng/mL
Arm/Group | Normal-BMI | Obese-MRI
Number analyzed (Participants) | 16 | 16
ng/mL | 18.2 [14.0 to 22.4] | 10.8 [6.8 to 14.8]

8. Secondary Outcome: Maximum Concentration of Serum UPA
Description: (Cmax) calculated in women with normal and obese BMI
Time Frame: Up to 24 hours
Measure: Mean (Inter-Quartile Range); unit: ng/mL
Arm/Group | Normal-BMI | Obese-MRI
Number analyzed (Participants) | 16 | 16
ng/mL | 89.3 [57.4 to 121.2] | 95.6 [65.8 to 125.4]

9. Secondary Outcome: Time to Maximum Concentration of Serum LNG
Description: (Tmax) calculated in women with normal and obese BMI
Time Frame: Up to 24 hours
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Normal-BMI | Obese-MRI
Number analyzed (Participants) | 16 | 16
h | 2.0 (2.0) | 3.0 (1.0)

10. Secondary Outcome: Time to Maximum Concentration of Serum UPA
Description: (Tmax) calculated in women with normal and obese BMI
Time Frame: Up to 24 hours
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Normal-BMI | Obese-MRI
Number analyzed (Participants) | 16 | 16
h | 1.6 (1.0) | 1.5 (1.0)

ADVERSE EVENTS:
Time Frame: 8 weeks
Description: The Total Number of Participants at Risk is not consistent with numbers provided in the rows in the Participant Flow module. There were 16 participants classified as "Normal-BMI" and 16 participants classified as "Obese-BMI", and all participants received all interventions; however, PRS instructed for the investigator to further split the 2 BMI arms into the time period when "Normal" and "Obese-BMI" received each drug, so that the reported events can be attributed to the appropriate drug.
Groups:
- Normal-BMI on LNG: Women with normal BMI will receive LNG-EC
- Normal-BMI on UPA; Obese-BMI on UPA: Women with obese BMI will receive UPA-EC
- Obese-BMI on LNG: Women with obese BMI will receive LNG-EC
Arm/Group | Normal-BMI on LNG | Normal-BMI on UPA | Obese-BMI on LNG | Obese-BMI on UPA
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 4/8 | 3/8 | 4/8 | 2/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Normal-BMI on LNG (N=8) | Normal-BMI on UPA (N=8) | Obese-BMI on LNG (N=8) | Obese-BMI on UPA (N=8)
Fatigue (General disorders) | 2 | 1 | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 2 | 0
Lower abdominal pain (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Pain (General disorders) | 1 | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No